CLINICAL TRIAL: NCT01173198
Title: A Prospective Evaluation of Outcomes Following Wavefront Optimized or Wavefront Guided Lasik Procedure in Low to Moderate Myopic Patients
Brief Title: An Evaluation of Outcomes Following Wavefront Optimized or Wavefront Guided Lasik Procedure in Low to Moderate Myopic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: David Schneider, MD, Midwest Eye Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WFG-002-WFO
Record Dates: First submitted 2010-02-01; First posted 2010-07-30 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Myopia
Keywords: LOW TO MODERATE MYOPIC PATIENTS
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WAVEFRONT GUIDED LASIK (Active Comparator)
  Interventions: Device: WAVEFRONT Optimized LASIK
- WAVEFRONT OPTIMIZED (Active Comparator)
  Interventions: Device: WAVEFRONT GUIDED LASIK

INTERVENTIONS:
Device: WAVEFRONT Optimized LASIK — 30 patients
  Arms: WAVEFRONT GUIDED LASIK
Device: WAVEFRONT GUIDED LASIK — 30 patients
  Arms: WAVEFRONT OPTIMIZED

SUMMARY:
To compare post-surgical outcomes in patients who have undergone Wavefront Guided LASIK (iLASIK platform) compared with patients who have undergone Wavefront Optimized LASIK (Wavelight Allegretto 400 Hz platform).

ELIGIBILITY:
Inclusion Criteria:

* The subject must be male or female, of any race, and at least 21 years old and not older than 35 years old at the time of the pre-operative examination;
* Both eyes must have a BSCVA of 20/20 or better;
* Both eyes must have a manifest refractive error from -2.00 D to -6.00 D, a cylinder component up to -1.50 D, and a maximum manifest spherical equivalent of -6.00 D;
* Both eyes must have at least 0.2 microns RMS HOA
* Both eyes must have a minimum pupil size of at least 6.0mm in dim illumination on wavescan;
* Both eyes must demonstrate refractive stability confirmed by clinical records or previous glasses. Refractive stability shall be documented by a change of less than or equal to 0.50 diopter (sphere and cylinder) at an exam at least 12 months prior to the baseline examination. The astigmatic axis must also be within 15 degrees for eyes with cylinder greater than 0.50 D; and
* Subjects should be willing and capable of returning for follow-up examinations for the duration of the study.

Exclusion Criteria:

* Use of systemic or ocular medications that may affect vision
* Subjects who use concurrent topical or systemic medications that may impair healing, including but not limited to: antimetabolites, isotretinoin (Accutane®) within 6 months of treatment, and amiodarone hydrochloride (Cordarone®) within 12 months of treatment; NOTE: The use of topical or systemic corticosteroids, whether chronic or acute, is deemed to adversely affect healing and subjects using such medication are specifically excluded from eligibility.
* Subjects with a history of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis; NOTE: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity or control, will specifically exclude subjects from eligibility.
* The subject must not have a history of prior intraocular or corneal surgery (including cataract extraction), active ophthalmic disease or abnormality (including, but not limited to, blepharitis, recurrent corneal erosion, dry eye syndrome, neovascularization > 1mm from limbus), clinically significant lens opacity, clinical evidence of trauma (including scarring), or with evidence of glaucoma or propensity for narrow angle glaucoma in either eye; NOTE: This includes any subject with open angle glaucoma, regardless of medication regimen or control.
* Subjects who have Amblyopia or strabismus
* Subjects with known pathology that may affect visual acuity; particularly retinal changes that affect vision (macular degeneration, cystoid macular edema, proliferative diabetic retinopathy, etc.)
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration, or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse
* Subjects who may be expected to require retinal laser treatment or other surgical intervention
* Subjects with pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 4.0 mm under mesopic/scotopic conditions)
* Contact lens usage within 6 months for PMMA contacts lenses, 1 month for gas permeable lenses or 1 week for extended-wear and daily-wear soft contact lenses
* Subject must not have any evidence of keratoconus, corneal irregularity, or abnormal videokeratography in either eye;
* Subjects with known sensitivity or inappropriate responsiveness to any of the medications used in the post-operative course;
* Patients who cannot obtain a Wavescan capture; and
* patients seeking monovision.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Reduction or elimination of myopia and myopic astigmatism | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Schneider, MD, Principal Investigator — MIdwest Eye Center
Locations (1):
- Midwest Eye Center, Cincinnati, Ohio, United States